CLINICAL TRIAL: NCT03197727
Title: Evaluation of Tooth Wear and Associated Risk Factors: a Matched Case-control Study
Brief Title: Tooth Wear and Associated Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Cansu Atalay, Postdoc reseacher, DDS, Ph.D, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GO14/519-01
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Tooth Wear
Keywords: Tooth wear, risk factors, saliva, diet, oral hygiene
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC Saliva-Check BUFFER (Other): Saliva test pH Buffering capacity Flow rate
  Interventions: Diagnostic Test: GC Saliva-Check BUFFER

INTERVENTIONS:
Diagnostic Test: GC Saliva-Check BUFFER — Evaluating the saliva flow rate, saliva pH and saliva buffering capacity

SUMMARY:
This study compares the associated risk factors between adults with tooth wear and age- and sex-matched controls without tooth wear.

DETAILED DESCRIPTION:
Some people are at greater risk due to their eating and brushing habits. Poor oral health behaviors and malnutrition are the leading causes of tooth surface loss in adults. Fluid consumption trends have changed, and the increased consumption of carbonated drinks coincides with a decline in the consumption of dairy products and increases in the use of packaged products. Frequent and faulty brushing with abrasive oral hygiene products can also increase TW. Individuals unhappy with the color of their teeth may also frequently use whitening toothpaste.

Saliva is considered the biological factor with the greatest potential to modify the progression of TW. There are several potential mechanisms by which saliva may protect enamel from dietary acid erosion. Saliva protection mechanisms include the dilution of erosive agents in the mouth, neutralization, effects of calcium and phosphate ions, and slowing of the rate of enamel dissolution.

The loss of dental tissue can lead to the character's loss of precision and form, and in advanced stages the dentin surface can be exposed. TW is initially painless and unrecognizable. In the next stage, complaints often include tenderness and non-aesthetic factors. It is difficult to recognize the signs of TW and very important to avoid premature diagnosis, as TW can often be diagnosed by a dentist. Correct diagnosis is an important part of the treatment and will help the dentist determine recommendations for the patient.

ELIGIBILITY:
Inclusion Criteria:

Subject is in good health. Subject is able to understand and read the questionnaire.

Exclusion Criteria:

Wearing orthodontic appliances, Having crowns or partial dentures Using any medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11-28 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2016-01-18 (Actual)

PRIMARY OUTCOMES:
Saliva test | 1 day
  Highly acidic saliva will be in the red section, pH 5.0 - 5.8. Moderately acidic saliva will be found in the yellow section, pH 6.0 - 6.6. Healthy saliva will be in the green section pH 6.8 - 7.8.

SECONDARY OUTCOMES:
Tooth wear | 1 day
  Scoring the tooth wear, Smith and Knight's index (0=No loss of enamel surface characteristics, 1=Loss of enamel surface characteristics, 2=Loss of enamel exposing dentine for less than one third of surface, 3=Loss of enamel exposing dentine for more than one third of the surface, 4=Complete enamel loss, pulp exposure, secondary dentine exposure

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fung A, Brearley Messer L. Tooth wear and associated risk factors in a sample of Australian primary school children. Aust Dent J. 2013 Jun;58(2):235-45. doi: 10.1111/adj.12055. Epub 2013 May 5. PMID 23713646
- [Background] El Aidi H, Bronkhorst EM, Huysmans MC, Truin GJ. Multifactorial analysis of factors associated with the incidence and progression of erosive tooth wear. Caries Res. 2011;45(3):303-12. doi: 10.1159/000328671. Epub 2011 Jun 8. PMID 21654171
- [Background] Zero DT, Lussi A. Erosion--chemical and biological factors of importance to the dental practitioner. Int Dent J. 2005;55(4 Suppl 1):285-90. doi: 10.1111/j.1875-595x.2005.tb00066.x. PMID 16167607